CLINICAL TRIAL: NCT04330573
Title: Sensory Characteristics and Psychosocial Factors Related With Non-specific Neck Musculoskeletal Pain Chronification
Acronym: CNSNP
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Collaborators: Hospital General de la Defensa en Zaragoza (Unknown)
Responsible Party: Principal Investigator, Pablo Herrero Gallego, Dr. Pablo Herrero, PT, PhD, Universidad San Jorge
Other Study IDs: CNSNP-USJ
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Neck Pain
Keywords: chronic non-specific neck pain; musculoskeletal pain; psychosocial factors; sensory characteristics; pressure pain thresholds; temporal summation
MeSH Terms: conditions — Neck Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Non-Specific Neck Pain: Patients with chronic non-specific neck pain. No interventions
  Interventions: Other: No intervention. Observational study
- Control/Healthy Group: Volunteers without pain. No interventions.
  Interventions: Other: No intervention. Observational study

INTERVENTIONS:
Other: No intervention. Observational study — Observational study

SUMMARY:
Chronic pain is commonly defined as any pain which lasts more than 12 weeks. Chronic non-specific neck pain (CNSNP) has no specific underlying disease causing the pain. There are neurophysiological factors that may modulate pain response and perception in the central nervous system, producing sensory changes such as the presence of temporal summation (TS) and pressure, cold or heat hyperalgesia. TS describes the progressive increase in reported pain intensity as a function of repeated noxious stimulation (e.g. thermal, electrical or mechanical). TS and hyperalgesia are measured through quantitative sensory tests (QST) where pain pressure thresholds (PPT) are measured with an algometer. The current evidence show that PPTs are significantly lower compared to healthy subjects and the association between PPTs, pain intensity and disability are inconsistent. Further, there are psychosocial factors (catastrophizing, kinesiophobia, stress…) that may influence the pain experience. This psychosocial factors associated with chronic pain are not systematically collected in the QST literature complicating the interpretation of data. The objectives of this study are 1) to determine disability, sensory (TS and PPTs) and psychosocial changes (kinesiophobia, catastrophizing, sleep quality, life quality, stress and anxiety) in the natural evolution or in the result of physiotherapy treatment in CNSNP individuals, 2) to study the correlations between disability, psychosocial and sensory factors and 3) to observe if there is a homogeneity between the subjects.

ELIGIBILITY:
Inclusion criteria for individuals with CNSNP were:

1. age between 18 and 65 years;
2. capable to understand, write, and speak in Spanish;
3. having suffered neck pain during the last 12 weeks at least;
4. pain localized in the neck region with or without pain radiation;
5. Negative Spurling test;
6. Negative Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS);
7. Negative Upper Limb Tension Test for the median nerve;
8. PainDetect test with non-neuropathic pain result. .

Exclusion Criteria:

1. Presence of red flag as reported in the medical history (i.e. tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis);
2. Neck pain with cervical radiculopathy;
3. fibromyalgia syndrome,
4. previous neck surgery;
5. currently undergoing any type of pain treatment or having received physical therapy in the previous 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was divided into 2 groups: individuals with Chronic Non-Specific Neck Pain and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index Change | T0 (baseline); T1 (1 month); T2 (6 months).
  It is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. Questions include activities of daily living, such as: personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration and headache. The 10 item scores are then summed to yield a global NDI score, which has a range of 0-50 where higher values reflect greater neck disability. 1 and 6-month results were subtracted from baseline. As such, positive change scores for neck disability indicate improvement
Quick-DASH change | T0 (baseline); T1 (1 month); T2 (6 months).
  The purpose of the QuickDASH is to use 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The QuickDASH is a widely used reference of self reported disability. The 11 item scores are then summed to yield a global QuickDASH score, which has a range of 11-100 where higher values reflect greater shoulder/arm disability. 1 and 6-month results were subtracted from baseline. As such, positive change scores for shoulder/arm disability indicate improvement

SECONDARY OUTCOMES:
Pressure Pain Threshold change | T0 (baseline); T1 (1 month); T2 (6 months).
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom.
Temporal Summation change | T0 (baseline); T1 (1 month); T2 (6 months).
  Temporal summation is a clinical measure of central sensitization in which a high frequency of action potentials in the presynaptic neuron elicits postsynaptic potentials that overlap and summate with each other.
Area of pain assessed by bodycharts change | T0 (baseline); T1 (1 month); T2 (6 months).
  Participants have to draw on a tablet-based digital body chart (NavigatePain©, Aalborg University, Aalborg, Denmark) the body region in which they felt pain more frequently during the previous month. The use of pain drawings has been found to be reliable in chronic low back, neck, shoulder, and arm pain. Digital pain drawings have also been shown reliable, valid and comparable to paper drawings and useful in clinical population. The size of the pain area was extracted and expressed in pixels.
Pain Intensity change- Visual Analogic Scale | T0 (baseline); T1 (1 month); T2 (6 months).
  Self-perceived neck pain will record using a Visual Analogue Scale (VAS). Participants have to mark on a 10-cm line their average current neck pain between 0 ("no pain") and 10 ("worst possible pain"). The VAS is a reliable and valid measurement of pain
Pain Duration change | T0 (baseline); T1 (1 month); T2 (6 months).
  Duration of pain in months
Catastrophism change. Pain Catastrophizing Scale | T0 (baseline); T1 (1 month); T2 (6 months).
  People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
Kinesiophobia change. Tampa Scale for Kinesiophobia | T0 (baseline); T1 (1 month); T2 (6 months).
  Tampa Scale for Kinesiophobia (TSK) The TSK is a 17-item self-report measure of fear of movement and (re)injury. Four of the items are negatively worded and reversed scored (4, 8, 12, and 16). Ratings are summed to yield a total score where higher values reflect greater fear of (re)injury. The 17 item scores are then summed to yield a global TSK score, which has a range of 11-44.
Quality of Life change. The 5-level EQ-5D version (EQ-5D-5L) | T0 (baseline); T1 (1 month); T2 (6 months).
  The EQ-5D is a frequently used generic quality of life questionnaire, designed by the EuroQoL. The EQ-5D-5L is an instrument widely used to measure and evaluate general health status. The EQ-5D-5L descriptive system describes general health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels, indicating no problems, slight problems, moderate problems, severe problems, and extreme problems resulting in a total of 3,125 unique health states. Besides, the EQ-5D-5L also includes a visual analogue scale (EQ-VAS), which recorded the patient's self-rated health on a 20 cm vertical, visual analogue scale with endpoints (0; 100) labeled 'the best health you can imagine' and 'the worst health you can imagine'
Stress change. Perceived Stress Scale | T0 (baseline); T1 (1 month); T2 (6 months).
  he Perceived Stress Scale (PSS) inquire about feelings and thoughts that tap the degree to which respondents find their current life situation unpredictable, uncontrollable and stressful. Respondents indicate how often in the past month they have felt or thought a certain way on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). The higher the score the higher the perceived stress is. The 14 item scores are then summed to yield a global PSS score, which has a range of 0-56
Quality of Sleep change . Pittsburgh Questionnaire | T0 (baseline); T1 (1 month); T2 (6 months).
  PSQI consists of 19 self-rated questions. The 19 self-rated questions asses a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep-related problems. Theses 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality.
Anxiety-Depression change. DASS 21. | T0 (baseline); T1 (1 month); T2 (6 months).
  The DASS is a self-report measure, designed to assess the unique and unrelated aspects of anxiety and depression, as well as a third construct (termed stress) that assesses the features common to anxiety and depression. The DASS-21 is comprised of three scales, Depression, Anxiety, and Stress, each of which consists of 7 items. The 21 item scores are then summed to yield a global DASS-21 score, which has a range of 0-63

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de la Defensa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be provided based on request to authors by email to gortego@usj.es